CLINICAL TRIAL: NCT05506956
Title: A Phase Ib to Investigate the CD123-targeted DART Flotetuzumab Following Allogeneic Transplant for Patients With CD123+ Acute Myeloid Leukemia
Brief Title: Post-transplant Flotetuzumab for AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: MacroGenics (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J21134; IRB00235421 (Other: JHMIRB); P01CA015396 (NIH)
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: CD123; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flotetuzumab Following Allogeneic Transplant (Experimental): All participants will receive one cycle (28 days) of flotetuzumab. After one cycle, all participants will undergo a bone marrow biopsy to assess response and based on the response, may receive additional cycles up to a total cycle of six cycles.
  Interventions: Drug: Flotetuzumab

INTERVENTIONS:
Drug: Flotetuzumab — Patients enrolled on dose level 1 (DL1) will receive flotetuzumab by continuous infusion using multi-step lead-in dosing, and then 500 ng/kg/day on days 7-28. After one cycle, all patients will undergo a bone marrow biopsy to assess response including assessment of minimal residual disease (MRD). Patients who fail to achieve a CR, CRi, CRh (complete remission with partial hematologic recovery), or MLFS may continue with subsequent induction cycles as a continuous infusion up to a total of five cycles. If there is evidence of response (CR, CRi, CRh, or MLFS) and the toxicities of treatment are acceptable, patients will be eligible for two consolidation cycles. Additional bone marrow biopsies for response assessment will be performed after the second cycle. If there is a need to de-escalate dosing based on toxicity, then patients will be enrolled on DL-1 using multi-step lead-in dosing, and then 300 ng/kg/day on days 5-28 of the first cycle and days 1-28 of subsequent cycles.

SUMMARY:
The purpose of this research study is to determine if the study drug, flotetuzumab, is safe and tolerable when given to participants with acute myeloid leukemia (AML) that has relapsed after transplant.

DETAILED DESCRIPTION:
Despite significant advances, the prognosis for patients with AML remains poor with 5-year overall survival of just ~40% in younger patients and much poorer long-term survival in older patients. Allogeneic hematopoietic stem cell transplantation (AlloHSCT) as post-remission therapy has led to improved overall survival when compared to consolidation chemotherapy for the vast majority of AML patients who have intermediate or poor risk cytogenetics. Due to significant transplant-related mortality (TRM) and poor outcomes in older patients with myeloablative conditioning (MAC) transplantation, there have been many studies investigating the feasibility of less intensive conditioning regimens such as reduced-intensity conditioning (RIC) and nonmyeloablative (NMA), which have shown comparable overall survival with decreased TRM but an increased risk of relapse. As these less intensive conditioning strategies become more widely adopted, the need to focus on the identification and treatment of AML patients at risk for post-transplant relapse increases. Maintenance therapy with tyrosine kinase inhibitors and monoclonal antibodies have proven safe and effective across a range of diseases including AML, acute lymphocytic leukemia (ALL), and non-Hodgkin's lymphoma (NHL). Leukemia stem cells (LSCs) are another potential target for post-transplant therapy, and the expression of CD123 readily discriminates AML LSCs from hematopoietic stem cells (HSCs). The anti-CD123 monoclonal antibody CSL360 has previously demonstrated efficacy in post-transplant patients with relapsed disease, while flotetuzumab has demonstrated efficacy in relapsed and refractory patients. Given this preliminary data, the investigators propose a trial of flotetuzumab as post-alloHSCT therapy for AML in patients with evidence of disease post-transplant including frank relapse. The investigators believe that treatment with flotetuzumab in this setting will be well tolerated and effective. Flotetuzumab is not approved for use in people with AML. Its use has not been specifically studied in patients with AML following a bone marrow transplant and therefore its use in this study is investigational.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed prior diagnosis of AML and underwent an alloHSCT as a form of consolidation in a morphologic complete remission
2. ECOG performance status 0-2
3. Ability to give informed consent
4. In agreement to use an effective barrier method of birth control to avoid pregnancy during the study and for a minimum of 30 days after study treatment, for all male and female patients who are fertile
5. Age ≥18 years
6. Prior treatment with a CD123-targeted therapy will be allowed assuming the patient did not have a grade 3 or 4 adverse reaction to prior use of this treatment
7. Normal thyroid function (defined by either a thyroid-stimulating hormone (TSH) within the reference range, a TSH above the reference range with a free T4 within the reference range, or a TSH below the reference range with both a free T4 and total T3 within the reference range) or normal thyroid tests on supplementation or treatment (defined as a TSH within the reference range)
8. Patients should be at least 30 days from transplant with morphologic evidence of disease progression on bone marrow biopsy
9. The presence of a CD123+ AML must be confirmed by flow cytometry with >1% CD123 AML blasts
10. Peripheral blast count ≤20,000/mm3 at time of initiation on Cycle 1 Day 1

Exclusion Criteria:

1. No evidence of donor engraftment (100% patient DNA in bone marrow or peripheral blood after alloHSCT based on either an unsorted specimen or CD3 sorted).
2. Active AML in central nervous system (CNS) or testes
3. Patients with active, uncontrolled infection. If an infection is controlled and under treatment, then the patient may become eligible.
4. Patients with active acute or chronic GVHD requiring GVHD therapy (mycophenolate mofetil, tacrolimus, sirolimus, or steroids) within 30 days
5. Patients without active acute or chronic GVHD requiring prophylactic GVHD therapy (mycophenolate mofetil, tacrolimus, sirolimus, or steroids) within 30 days
6. Inadequate end organ function defined as:

   * Hepatic-AST, ALT, and alkaline phosphatase > 3.5X upper limit of normal (ULN), bilirubin >2.5X ULN
   * Renal-creatinine clearance <60 mL/min using the modified Cockcroft-Gault formula
   * Cardiac-Recent myocardial infarction within 6 months, Congestive Heart Failure with ejection fraction (EF) <50%, active pericarditis or myocarditis
   * Pulmonary-Need for supplemental oxygen to maintain oxygen saturation >92%
   * Adrenal-Adrenal insufficiency requiring physiologically-dosed steroids
7. Women who are pregnant or lactating
8. Previous or known hypersensitivity to biological agents or constituents of flotetuzumab or its source material
9. Concurrent use of any other investigational drugs
10. Uncontrolled infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus (HCV)
11. Any active untreated autoimmune disorders (with the exception of vitiligo, resolved childhood atopic dermatitis, prior Grave's disease now euthyroid clinically with stable supplementation)
12. Previous treatment with radiotherapy or an immunotherapeutic agent in the 14 days prior to study drug administration (Cycle 1 Day 1) or 5 half-lifes, whichever is longer
13. Requirement, at the time of study entry, for concurrent steroids > 10 mg/day of oral prednisone or equivalent, except steroid inhaler, nasal spray, or ophthalmic solution
14. Use of granulocyte colony stimulating or granulocyte-macrophage colony stimulating factor in the 2 weeks prior to study drug administration
15. Prior adverse event with CD123 therapy necessitating therapy discontinuation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Webster, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants receive dose level 1 (DL1): Flotetuzumab: 500 ng/kg/day. No participants received DL-1: Flotetuzumab: 300 ng/kg/day during the study.
Groups:
- Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day: All participants will receive one cycle (28 days) of flotetuzumab. After one cycle, all participants will undergo a bone marrow biopsy to assess response and based on the response, may receive additional cycles up to a total cycle of six cycles.
  Flotetuzumab: Patients enrolled on dose level 1 (DL1) will receive flotetuzumab by continuous infusion using multi-step lead-in dosing, and then 500 ng/kg/day on days 7-28. After one cycle, all patients will undergo a bone marrow biopsy to assess response including assessment of minimal residual disease (MRD). Patients who fail to achieve a CR, CRi, CRh (complete remission with partial hematologic recovery), or MLFS may continue with subsequent induction cycles as a continuous infusion up to a total of five cycles. If there is evidence of response (CR, CRi, CRh, or MLFS) and the toxicities of treatment are acceptable, patients will be eligible for two consolidation cycles. Additional bone marrow biopsies for response assessment will be performed after the second cycle.
  If there is a need to de-escalate dosing based on toxicity, then patients will be enrolled on DL-1 using multi-step lead-in dosing, and then 300 ng/kg/day on days 5-28 of the first cycle and days 1-28 of subsequent cycles.
Period: Overall Study
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 69 [63 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities to Determine Maximum Tolerated Dose (MTD) of Flotetuzumab in Patients With Relapsed/Refractory AML Following alloHSCT
Description: Number of participants with dose-limiting toxicities (DLTs) at specified dose levels to determine MTD
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day: Multi-step lead-in dosing on days 1-7 followed by 500 ng/kg/day on days 7-28
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Complete Response to Flotetuzumab in Patients With Relapsed AML Following Allogeneic Hematopoietic Stem Cell Transplant (alloHSCT)
Description: Number of participants with complete response (CR) following alloHSCT.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Complete Response With Incomplete Count Recovery to Flotetuzumab in Patients With Relapsed AML Following alloHSCT
Description: Number of participants with complete response with incomplete count recovery (CRi) following allogeneic hematopoietic stem cell transplant (alloHSCT).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Partial Response to Flotetuzumab in Patients With Relapsed AML Following alloHSCT
Description: Number of participants with partial response (PR) following allogeneic hematopoietic stem cell transplant (alloHSCT).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Acute Graft-versus-host Disease (GVHD) Incidence
Description: Number of safety events defined as CTCAE grade III-IV acute GVHD.
Time Frame: 6 months
Measure: Number; unit: events
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
events | 0

6. Secondary Outcome: Chronic GVHD Incidence
Description: Number of events of chronic GVHD requiring systemic immune suppression
Time Frame: 6 months
Measure: Number; unit: events
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
events | 0

7. Secondary Outcome: Non-relapse Mortality
Description: Number of participant deaths without recurrent or progressive disease after allo-HSCT.
Time Frame: through study completion, an average of 1 year 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, approximately 1 year 8 months
Arm/Group | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day (N=3)
Cytokine Release Syndrome (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (DL1): Flotetuzumab: 500 ng/kg/Day (N=3)
Fever (Immune system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT05506956/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT05506956/ICF_001.pdf